CLINICAL TRIAL: NCT03049319
Title: Comparing Minimal Erythema Dose (MED) in UVB Devices in the Presence and Absence of UV Filter
Brief Title: MED in UVB Devices in the Presence and Absence of UV Filter
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor did not provide the equipment needed to do study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00042226
Record Dates: First submitted 2017-02-07; First posted 2017-02-10 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Healthy Participants and/or Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Laser (Experimental): All six interventions will be applied to patient's back.
  Interventions: Device: Psoriashield in the presence of a non-UV absorbing block.; Device: Psoriashield in the presence of a UV absorbing block.; Device: Psoriashield; Device: Xtrac laser in the presence of a non-UV absorbing block.; Device: Xtrac in the presence of a UV absorbing block.; Device: Xtrac laser

INTERVENTIONS:
Device: Psoriashield in the presence of a non-UV absorbing block. — The psoriashield will be applied to patient's back in the presence of a non-UV absorbing block.
Device: Psoriashield in the presence of a UV absorbing block. — The psoriashield will be applied to patient's back in the presence of a UV absorbing block.
Device: Psoriashield — The psoriashield will be applied to patient's back.
Device: Xtrac laser in the presence of a non-UV absorbing block. — The Xtrac laser will be applied to patient's back in the presence of a UV absorbing block.
Device: Xtrac in the presence of a UV absorbing block. — The Xtrac laser will be applied to patient's back in the presence of a non-UV absorbing block.
Device: Xtrac laser — The Xtrac laser will be applied to patient's back.

SUMMARY:
Psoriasis affects 2-3% of the American population. While a wide variety of therapies currently exist, including topical corticosteroids and Vit D analogs, oral immunosuppressant and retinoid agents a better understanding of phototherapy is needed. Given the prevalence of localized psoriasis and dissatisfaction with treatment, investigation of localized treatment should be a priority for researchers with goals to improve the current standard of care.

DETAILED DESCRIPTION:
Psoriasis affects 2-3% of the American population. Psoriasis involving less than 10% BSA in the absence of joint involvement tends to be treated locally. More than 80% of people with psoriasis have <10% BSA involvement. A wide variety of therapies currently exist, including topical corticosteroids and Vit D analogs, oral immunosuppressant, retinoid agents, and phototherapy. Given the prevalence of localized psoriasis and dissatisfaction with treatment, investigation of localized treatment should be a priority for researchers with goals to improve the current standard of care.

UV light has a wavelength of 10nm - 380nm, which is slightly shorter than the wavelength of visible light. The UV light can be further classified to a narrow spectrum (UVB light has a wavelength of 280-315 nm). UVA has a wavelength of 315-400nm. Tanning beds use UV light to produce their effects. Whole body ultraviolet B (UVB) phototherapy is efficacious and is recommended as a first line option in selective psoriasis treatment recommendations. In pregnancy, UVB therapy is recommended as first line treatment for extensive plaque and guttate psoriasis.

Although UVB phototherapy has been included in the guidelines for psoriasis treatment, its use does not come without risk. Toxicities include cataract formation, herpes reactivation, photoaging, and with long-term exposure may lead to an increased risk of genital tumors in males. In addition, the use of UVB is rarely used as a first-line treatment for localized psoriasis probably due to financial issues and increased requirements for clinic visits. Narrowband UVB therapy (emission 311- 313nm) is superior to broad-band UVB light, and reduces toxicity. Psoriatic plaques can withstand much higher doses of UV light than the surrounding uninvolved skin; UV treatment of just the involved skin therefore offers increased efficacy in fewer treatments. In addition, localized treatment may remain in remission even 4 months after clearing with localized laser treatment. Localized treatment should therefore be a more favorable treatment option for psoriasis, using higher doses with sparing of healthy skin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 18 years of age.
* Good health as determined by lack of clinically significant abnormalities in medical history and clinical assessment, as judged by the Investigator.
* Subject is capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* The subject is able to complete the study and comply with study instructions, including attending all study visits.
* If a female subject of childbearing potential, subject has a negative urine pregnancy test.

Exclusion Criteria:

* Subject has a history of being non-responsive to UVB therapy
* Subject received phototherapy in the past four weeks
* Subject used topical therapy within two weeks from baseline (Excluding emollients)
* Subject has used experimental drugs or devices at least one month prior to Baseline
* Subject has a known history of Photosensitivity disorder (Including Xeroderma pigmentosum, SLE, Cockayne Syndrome, Bloom Syndrome) or is currently taking any medication that causes photosensitivity that requires they avoid sunlight.
* Subject has other serious skin disorder or any chronic medical condition that is not well controlled.
* Subject has major illness within 30 days prior to the Baseline visit.
* Subject has history of any immunocompromising disease.
* Subject is pregnant or nursing. Pregnant and nursing females will not be allowed in the study, and females of childbearing potential will have a pregnancy test at Baseline.
* Subject has a skin condition or disease that may require concurrent therapy or may confound the evaluation.
* Presence of any skin condition or coloration that would interfere with placement of test sites or the response or assessment of MED.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
MED Reading | 24 hours
  Minimal Erythemal Dose

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Elias Oussedik, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feldman SR, Mellen BG, Housman TS, Fitzpatrick RE, Geronemus RG, Friedman PM, Vasily DB, Morison WL. Efficacy of the 308-nm excimer laser for treatment of psoriasis: results of a multicenter study. J Am Acad Dermatol. 2002 Jun;46(6):900-6. doi: 10.1067/mjd.2002.120454. PMID 12063488
- [Background] Walters IB, Burack LH, Coven TR, Gilleaudeau P, Krueger JG. Suberythemogenic narrow-band UVB is markedly more effective than conventional UVB in treatment of psoriasis vulgaris. J Am Acad Dermatol. 1999 Jun;40(6 Pt 1):893-900. doi: 10.1016/s0190-9622(99)70076-9. PMID 10365919